CLINICAL TRIAL: NCT00002589
Title: Adjuvant Autolymphocyte Therapy (ALT) For Patients With Non-Metastatic Renal Cell Carcinoma
Brief Title: Lymphocyte Therapy in Treating Patients With Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000063744; STLMC-BRM-9401; NCI-V94-0514
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-12

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Muromonab-CD3; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: muromonab-CD3
Biological: therapeutic autologous lymphocytes
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Treating a person's lymphocytes with interleukin-2 and monoclonal antibody may help them kill more cancer cells when they are put back in the body.

PURPOSE: This phase II trial is studying how well lymphocyte therapy works in treating patients with stage III or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the ability of autologous lymphocyte therapy (ALT) given as adjuvant therapy following nephrectomy and/or complete surgical resection of any metastatic disease to delay or prevent metastatic recurrence in patients with high-risk renal cell carcinoma.
* Determine the incidence of tumor recurrence and the survival of these patients treated with this regimen.
* Determine the toxicity/morbidity of this regimen in these patients.
* Explore the relationship between clinical response and in vitro autologous lymphocyte characteristics, including lytic activity, cytokine production, response to cytokines, and phenotypic profile in these patients treated with this regimen.
* Assess patient immune status before, during, and after therapy.

OUTLINE: Patients are stratified according to postnephrectomy interval (less than 3 months vs more than 3 months), extent of lymph node involvement (N1 vs N2-N3), interleukin-1 concentration in initial autologous lymphocyte culture (less than 500 pg/mL vs greater than 500 pg/mL), and prenephrectomy treatment.

Mononuclear cells are collected by apheresis on day 1 and cultured with interleukin-2 and monoclonal antibody OKT3. After cellular production, the autologous lymphocytes are reinfused over at least 30 minutes. Treatment repeats monthly for 6 months and then every 3 months for 6 months in the absence of unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 10-90 patients will accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented and completely resected stage III or stage IV renal cell carcinoma, clinically staged within 2 months prior to initiation of therapy
* No evidence of nephrotic syndrome

PATIENT CHARACTERISTICS:

Age:

* Over 16

Performance status:

* ECOG 0-2

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count 50,000/mm3 to 500,000/mm^3
* Hemoglobin at least 10 g/dL
* No hematologic abnormalities

Hepatic:

* PT no greater than 1.5 times control
* PTT less than 1.5 times control
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 4.0 mg/dL
* Calcium no greater than 12 mg/dL
* No symptomatic hypercalcemia

Cardiovascular:

* No uncontrolled or severe cardiac disease, e.g.:

  * No myocardial infarction within 6 months
  * No congestive heart failure

Other:

* HIV negative
* No significant organ dysfunction
* No other serious medical illness that would limit life expectancy
* No significant CNS disease including uncontrolled or untreated psychiatric or seizure disorders
* No uncontrolled bacterial, viral, or fungal infection
* No active peptic or duodenal ulcer
* Adequate peripheral venous access required
* No prior malignancy within past 5 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* No other concurrent postnephrectomy adjuvant therapy

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* More than 1 week since prior corticosteroids (except as inhalation therapy for respiratory ailments or replacement for adrenal insufficiency)
* No concurrent therapy with the following:

  * Estrogens (except as postmenopausal replacement therapy)
  * Androgens
  * Progestins
  * Antiestrogens
  * Antiandrogens
  * LHRH analogues or antagonists
  * Other hormones

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No prior solid organ allograft
* More than 3 weeks since major surgery, including nephrectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 1994-07

PRIMARY OUTCOMES:
Survival as measured by Kaplan-Meier method at 5 years
Onset of recurrence as measured by Kaplan-Meier method at 5 years
Safety as measured by NCI Common Toxicity Criteria at completion of study

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States